CLINICAL TRIAL: NCT00511589
Title: PCR in Blood Cultures of Individuals With Positive and Inconclusive Serology for Chagas' Disease
Brief Title: Chagas Disease Diagnostic - Inconclusive Serology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Model: Parallel | Masking: None
Other Study IDs: upeclin/HC/FMB-Unesp-pre01
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2007-08

CONDITIONS: Parasitemia; Protozoan Infections
MeSH Terms: conditions — Parasitemia; Protozoan Infections

INTERVENTIONS:
Other: chagas disease diagnostic

SUMMARY:
T. cruzi infection affects approximately five million people in Brazil. The diagnosis of the chronic phase of infection is performed by indirect serological methods which, nevertheless, leave inconclusive results. One of the direct methods used for T. cruzi identification, blood culture in LIT (liver infusion tryptose) medium, presents low sensitivity in that phase of the disease. A negative result does not eliminate the possibility of infection, but a positive test has high absolute diagnostic value, which enables the indication of antiparasitic treatment. Molecular diagnosis (PCR) in this phase is promising and can be used as a confirmatory test, particularly when individuals present inconclusive results in conventional serological tests, such as ELISA, HAI and IFI. This study aimed at improving blood culture sensitivity in LIT medium by performing PCR in individuals with positive and inconclusive serology for chagasic infection.

ELIGIBILITY:
Inclusion Criteria:

* individuals with positive or inconclusive results in conventional serological tests: ELISA, HAI and IFI for Chagas disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Mariele Cristina M Picka, MSc, Principal Investigator — UPECLIN HC FM Botucatu Unesp
Locations (1):
- Univerdidade Estadual Paulista, Botucatu, São Paulo, Brazil